CLINICAL TRIAL: NCT03351231
Title: A Phase 1/2a Study of BMS-986242 Administered in Combination With Nivolumab (BMS-936558, Anti-PD-1) in Advanced Malignant Tumors
Brief Title: An Investigational Immuno-Therapy Study of Experimental Medication BMS-986242 Given in Combination With Nivolumab in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to meet protocol objectives
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA024-001; 2017-003603-21 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab; spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): BMS-986242 administered in combination with Nivolumab
  Interventions: Drug: BMS-986242; Biological: Nivolumab
- Dose Expansion (Experimental): BMS-986242 administered in combination with Nivolumab
  Interventions: Drug: BMS-986242; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986242 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Anti-PD-1

SUMMARY:
The purpose of this study is to investigate safety of experimental medication BMS-986242 and Nivolumab in patients with advanced cancers.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologic or cytological confirmation of a malignancy that is advanced (metastatic and/or unresectable) with measureable disease per RECIST v1.1
* Participants must have received and then progressed or been intolerant to at least 1 standard treatment regimen in the advanced or metastatic setting if such a therapy exists
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Ability to swallow tablets
* Adequate bone marrow and organ function, as defined by the protocol

Exclusion Criteria:

* Participants with known or suspected CNS metastases, untreated CNS metastases, or with the CNS as the only site of disease (patients with controlled brain metastasis allowed to enroll)
* Ocular melanoma
* Any significant acute or chronic medical illness
* Prior malignancy
* Other active malignancy requiring concurrent intervention
* Prior organ allograft or allogeneic bone marrow transplantation
* Participants with active, known, or suspected autoimmune disease
* Requirement for daily supplemental oxygen
* Uncontrolled or significant cardiovascular disease
* Pre-existing liver disease
* Gastrointestinal disease known to interfere with absorption

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Hoag Memorial Hospital Presbyterian, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Local Institution, Baltimore, Maryland

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were enrolled and 5 of those participants entered treatment; reasons for 2 participants not entering treatment were due to: 1 death; 1 participant no longer met study criteria. Note: study terminated following starting dose of BMS-986242 12.5 mg; dosing did not escalate.
Groups:
- BMS-986242 12.5 mg + Nivolumab 480 mg: 2-week monotherapy of BMS986-242 (Cycle 0), followed by combination treatment cycles every 4 weeks for 104 weeks (or 26 cycles); each treatment cycle consists of daily oral dose of BMS-986242 and 1 dose of Nivolumab intravenously every 4 weeks on Day 1 of treatment cycle; every 2 treatment cycles decision may be made to add cycles of study treatment based on radiological tumor assessments
Period: Combination Therapy Period
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Started | 5 (Started = initiated and completed monotherapy, then initiated combination therapy)
Completed | 0 (Completed = finished combination therapy)
Not Completed | 5
Not completed — Administrative reason by the Sponsor | 1
Not completed — Disease progression | 2
Not completed — Study drug toxicity | 1
Not completed — Adverse Event unrelated to study drug | 1
Period: Safety Follow-Up Period
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Started | 3 (Started = Initiated Safety Follow-up)
Completed | 0 (Completed = Finishing safety follow-up and continuing in study)
Not Completed | 3
Not completed — Participant withdrew consent | 1
Not completed — Other reason | 2

BASELINE CHARACTERISTICS:
Population: All treated participants; Note: study terminated following starting dose of BMS-986242 12.5 mg; dosing did not escalate.
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: The primary objective to establish safety to be measured by the primary endpoint of AEs
Time Frame: From initiation of study treatment until 100 days after discontinuation of study treatment
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of participants | NA — Study terminated, data not reported due to privacy reasons

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: The primary objective to establish safety to be measured by the primary endpoint of SAEs
Time Frame: From the date of participant's written consent until 100 days after discontinuation of nivolumab or participation in the study
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of participants | NA — Study terminated, data not reported due to privacy reasons

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: The primary objective to establish safety to be measured by the primary endpoint of dose limiting toxicities
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of participants | NA — Study terminated, data not reported due to privacy reasons

4. Primary Outcome: Number of Participants With AEs Leading to Discontinuation
Description: The primary objective to establish safety to be measured by the primary endpoint of AEs leading to discontinuation
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of participants | NA — Study terminated, data not reported due to privacy reasons

5. Primary Outcome: Number of Deaths
Description: The primary objective to establish safety to be measured by the primary endpoint of deaths
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of deaths
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of deaths | NA — Study terminated, data not reported due to privacy reasons

6. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: The primary objective to establish safety to be measured by the primary endpoint of clinical laboratory test abnormalities
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 5
Number of participants | NA — Study terminated, data not reported due to privacy reasons

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Pharmacokinetic (PK) parameters are assessed for BMS-986242 and selected metabolites following single-dose administration in Cycle 00 and multiple-dose administration in Cycle 0
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

9. Secondary Outcome: Area Under the Concentration-time Curve in 1 Dosing Interval [AUC(TAU)]
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity [AUC(INF)]
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Trough Observed Plasma Concentration at the End of the Dosing Interval (Ctrough)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Apparent Elimination Half-life (T-HALF)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: Apparent Total Body Clearance (CLT/F)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

15. Secondary Outcome: Accumulation Index (AI)
Description: The Pharmacokinetic (PK) parameters are assessed for BMS-986242 and selected metabolites following single-dose administration in Cycle 00 and multiple-dose administration in Cycle 0.
  Accumulation index, calculated based on ratio of area under the curve (AUC) and Cmax at steady state to after the first dose.
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

16. Secondary Outcome: Percent Urinary Recovery Over 24 Hours (%UR24)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

17. Secondary Outcome: Percent Urinary Recovery Over 72 Hours (%UR72)
Description: as for outcome 7
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

18. Secondary Outcome: Incidence of Anti-drug Antibody (ADA) to Nivolumab in Combination With BMS-986242
Description: Baseline ADA-positive participant is defined as a participant who has a ADA detected sample at baseline. ADA-positive participant is a participant with at least 1 ADA-positive sample relative to baseline after initiation of the treatment.
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

19. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR in participants with a best overall response (BOR) of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for solid tumors
Time Frame: Approximately 2 years
Population: Study terminated, data not reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are monitored from initiation of study treatment (monitored from participant's written consent for Serious Adverse Events) up through 100 days post-End of Treatment (EOT); Study Start of December 2017 and Study End of August 2018 (assessed approximately 1 year)
Description: The study will not be reported due to privacy reasons
Arm/Group | BMS-986242 12.5 mg + Nivolumab 480 mg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT03351231/Prot_SAP_000.pdf